CLINICAL TRIAL: NCT02136134
Title: Phase 3 Study Comparing Daratumumab, Bortezomib and Dexamethasone (DVd) vs Bortezomib and Dexamethasone (Vd) in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Addition of Daratumumab to Combination of Bortezomib and Dexamethasone in Participants With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR103995; 2014-000255-85 (EudraCT Number); 54767414MMY3004 (Other: Janssen Research & Development, LLC); NCT01620879 (obsolete NCT alias)
Record Dates: First submitted 2014-05-01; First posted 2014-05-12 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Plasmacytoma; Refractory Multiple Myeloma; Relapsed Multiple Myeloma; Daratumumab; VELCADE
MeSH Terms: conditions — Multiple Myeloma; Plasmacytoma | interventions — daratumumab; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daratumumab+VELCADE+dexamethasone (Experimental): Daratumumab, VELCADE and dexamethasone
  Interventions: Drug: Daratumumab; Drug: VELCADE (Bortezomib); Drug: Dexamethasone
- VELCADE+dexamethasone (Active Comparator): VELCADE and dexamethasone.
  Interventions: Drug: VELCADE (Bortezomib); Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Daratumumab will be administered as an IV infusion or 16 mg/kg weekly for the first 3 cycles, on Day 1 of Cycles 4-9, and then every 4 weeks thereafter. As per protocol amendment-6 participants receiving treatment with daratumumab IV will have the option to switch to daratumumab SC 1800 mg on Day 1 of any cycle, at the discretion of the investigator.
  Arms: Daratumumab+VELCADE+dexamethasone
Drug: VELCADE (Bortezomib) — VELCADE will be administered at a dose of 1.3 mg/m2 subcutaneously (SC) on Days 1, 4, 8 and 11 of each 21-day cycle. Eight VELCADE treatment cycles are to be administered.
  Other Names: VELCADE
Drug: Dexamethasone — Dexamethasone will be administered orally at 20 mg on Days 1, 2, 4, 5, 8, 9, 11 and 12 of the first 8 VELCADE treatment cycles.

SUMMARY:
The purpose of this study is to assess the effects of administration of daratumumab when combined with VELCADE (bortezomib) and dexamethasone compared with bortezomib and dexamethasone alone, for participants with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
This is an open-label (physicians and participants know the identity of the assigned treatment), randomized (the study medication is assigned by chance), multicenter, active-controlled study comparing daratumumab, VELCADE, and dexamethasone (DVd) with VELCADE and dexamethasone (Vd) in participants with relapsed or refractory multiple myeloma. Approximately 480 participants will be randomly assigned in a 1:1 ratio to receive either DVd or Vd. Randomization will be stratified by International Staging System (ISS), number of prior treatment programs (1 vs. 2 or 3 vs. >3), and prior VELCADE treatment ("no" vs. "yes"). Within each stratum, participants will be randomized to one of the treatment groups.The study will consist of a Screening Phase, a Treatment Phase, and a Follow-up Phase. Participants will be treated until disease progression, unacceptable toxicity, or other reasons to discontinue the study.

ELIGIBILITY:
Inclusion Criteria:

* Must have had documented multiple myeloma
* Must have received at least 1 prior line of therapy for multiple myeloma
* Must have had documented evidence of progressive disease as defined based on Investigator's determination of response of International Myeloma Working Group (IMWG) criteria on or after their last regimen
* Must have an Eastern Cooperative Oncology Group Performance Status score of 0, 1, or 2
* Must have achieved a response (partial response [PR] or better based on investigator's determination of response by the IMWG criteria) to at least 1 prior regimen in the past

Exclusion Criteria:

* Has received daratumumab or other anti-CD38 therapies previously
* Is refractory to VELCADE or another PI, like ixazomib and carfilzomib (had progression of disease while receiving VELCADE therapy or within 60 days of ending VELCADE therapy or another PI therapy, like ixazomib and carfilzomib
* Is intolerant to VELCADE (ie, discontinued due to any adverse event while on VELCADE treatment)
* Has received anti-myeloma treatment within 2 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is longer, before the date of randomization. The only exception is emergency use of a short course of corticosteroids (equivalent of dexamethasone 40 milligram per day [mg/day] for a maximum of 4 days) before treatment. A list of anti-myeloma treatments with the corresponding pharmacokinetic half-lives is provided in the Site Investigational Product Procedures Manual (IPPM).
* Has a history of malignancy (other than multiple myeloma) within 3 years before the date of randomization
* Has any concurrent medical condition or disease (eg, active systemic infection) that is likely to interfere with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2014-08-15 (Actual); Primary Completion 2016-01-11 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical trial, Study Director — Janssen Research & Development, LLC
Locations (105):
- United States (17):
  - Birmingham, Alabama
  - Los Angeles, California
  - Stamford, Connecticut
  - Jacksonville, Florida
  - Atlanta, Georgia
  - Niles, Illinois
  - Topeka, Kansas
  - Westwood, Kansas
  - Marrero, Louisiana
  - Boston, Massachusetts
  - Lansing, Michigan
  - New York, New York
  - Chapel Hill, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Seattle, Washington
- Australia (7):
  - Adelaide
  - Concord
  - Fitzroy
  - Hobart
  - Melbourne
  - Nedlands
  - Woodville South
- Brazil (4):
  - Barretos
  - Porto Alegre
  - Salvador
  - São Paulo
- Czechia (4):
  - Brno
  - Hradec Králové
  - Ostrava-Poruba
  - Prague
- Germany (12):
  - Bamberg
  - Berlin
  - Düsseldorf
  - Freiburg im Breisgau
  - Göttingen
  - Hamburg
  - Mainz
  - München
  - Stuttgart
  - Tübingen
  - Ulm
  - Würzburg
- Hungary (5):
  - Budapest
  - Debrecen
  - Győr
  - Pécs
  - Veszprém
- Mexico (2):
  - Huixquilucan
  - Monterrey
- Netherlands (8):
  - Alkmaar
  - Amersfoort
  - Dordrecht
  - Groningen
  - Leiden
  - Maastricht
  - Nijmegen
  - The Hague
- Poland (5):
  - Chorzów
  - Katowice
  - Krakow
  - Poznan
  - Warsaw
- Russia (9):
  - Krasnodar
  - Moscow
  - Nizhny Novgorod
  - Penza
  - Pyatigorsk
  - Ryazan
  - Samara
  - Sochi
  - Syktyvkar
- South Korea (5):
  - Busan
  - Hwasun
  - Seoul
  - Suwon
  - Ulsan
- Spain (5):
  - Madrid
  - Salamanca
  - San Sebastián de los Reyes
  - Toledo
  - Valencia
- Sweden (8):
  - Linköping
  - Luleå
  - Lund
  - Örebro
  - Sundsvall
  - Umeå
  - Uppsala
  - Västerås
- Turkey (Türkiye) (6):
  - Ankara
  - Istanbul
  - Izmir
  - Kayseri
  - Kocaeli
  - Malatya
- Ukraine (8):
  - Cherkasy
  - Dnipro
  - Ivano-Frankivsk
  - Kiev
  - Lviv
  - Poltava
  - Vinnitsa
  - Zaporizhzhya

REFERENCES:
- [Derived] Almansour SA, Alqudah MAY, Abuhelwa Z, Al-Shamsi HO, Alhuraiji A, Semreen MH, Bustanji Y, Alzoubi KH, Modi ND, Mckinnon RA, Sorich MJ, Hopkins AM, Abuhelwa AY. Antithrombotic utilization, adverse events, and associations with treatment outcomes in multiple myeloma: pooled analysis of three clinical trials. Ther Adv Med Oncol. 2024 Sep 2;16:17588359241275387. doi: 10.1177/17588359241275387. eCollection 2024. PMID 39229471
- [Derived] Spencer A, Moreau P, Mateos MV, Goldschmidt H, Suzuki K, Levin MD, Sonneveld P, Orlowski RZ, Yoon SS, Usmani SZ, Weisel K, Reece D, Ahmadi T, Pei H, Mayo WG, Gai X, Carey J, Bartlett JB, Carson R, Dimopoulos MA. Daratumumab for patients with myeloma with early or late relapse after initial therapy: subgroup analysis of CASTOR and POLLUX. Blood Adv. 2024 Jan 23;8(2):388-398. doi: 10.1182/bloodadvances.2023010579. PMID 38048391
- [Derived] Sonneveld P, Chanan-Khan A, Weisel K, Nooka AK, Masszi T, Beksac M, Spicka I, Hungria V, Munder M, Mateos MV, Mark TM, Levin MD, Ahmadi T, Qin X, Garvin Mayo W, Gai X, Carey J, Carson R, Spencer A. Overall Survival With Daratumumab, Bortezomib, and Dexamethasone in Previously Treated Multiple Myeloma (CASTOR): A Randomized, Open-Label, Phase III Trial. J Clin Oncol. 2023 Mar 10;41(8):1600-1609. doi: 10.1200/JCO.21.02734. Epub 2022 Nov 22. PMID 36413710
- [Derived] He J, Berringer H, Heeg B, Ruan H, Kampfenkel T, Dwarakanathan HR, Johnston S, Mendes J, Lam A, Bathija S, Mackay EK. Indirect Treatment Comparison of Daratumumab, Pomalidomide, and Dexamethasone Versus Standard of Care in Patients with Difficult-to-Treat Relapsed/Refractory Multiple Myeloma. Adv Ther. 2022 Sep;39(9):4230-4249. doi: 10.1007/s12325-022-02226-x. Epub 2022 Jul 22. PMID 35876974
- [Derived] Cavo M, San-Miguel J, Usmani SZ, Weisel K, Dimopoulos MA, Avet-Loiseau H, Paiva B, Bahlis NJ, Plesner T, Hungria V, Moreau P, Mateos MV, Perrot A, Iida S, Facon T, Kumar S, van de Donk NWCJ, Sonneveld P, Spencer A, Krevvata M, Heuck C, Wang J, Ukropec J, Kobos R, Sun S, Qi M, Munshi N. Prognostic value of minimal residual disease negativity in myeloma: combined analysis of POLLUX, CASTOR, ALCYONE, and MAIA. Blood. 2022 Feb 10;139(6):835-844. doi: 10.1182/blood.2021011101. PMID 34289038
- [Derived] Avet-Loiseau H, San-Miguel J, Casneuf T, Iida S, Lonial S, Usmani SZ, Spencer A, Moreau P, Plesner T, Weisel K, Ukropec J, Chiu C, Trivedi S, Amin H, Krevvata M, Ramaswami P, Qin X, Qi M, Sun S, Qi M, Kobos R, Bahlis NJ. Evaluation of Sustained Minimal Residual Disease Negativity With Daratumumab-Combination Regimens in Relapsed and/or Refractory Multiple Myeloma: Analysis of POLLUX and CASTOR. J Clin Oncol. 2021 Apr 1;39(10):1139-1149. doi: 10.1200/JCO.20.01814. Epub 2021 Jan 29. PMID 33513030
- [Derived] Weisel K, Spencer A, Lentzsch S, Avet-Loiseau H, Mark TM, Spicka I, Masszi T, Lauri B, Levin MD, Bosi A, Hungria V, Cavo M, Lee JJ, Nooka A, Quach H, Munder M, Lee C, Barreto W, Corradini P, Min CK, Chanan-Khan AA, Horvath N, Capra M, Beksac M, Ovilla R, Jo JC, Shin HJ, Sonneveld P, Casneuf T, DeAngelis N, Amin H, Ukropec J, Kobos R, Mateos MV. Daratumumab, bortezomib, and dexamethasone in relapsed or refractory multiple myeloma: subgroup analysis of CASTOR based on cytogenetic risk. J Hematol Oncol. 2020 Aug 20;13(1):115. doi: 10.1186/s13045-020-00948-5. PMID 32819447
- [Derived] Mateos MV, Spencer A, Nooka AK, Pour L, Weisel K, Cavo M, Laubach JP, Cook G, Iida S, Benboubker L, Usmani SZ, Yoon SS, Bahlis NJ, Chiu C, Ukropec J, Schecter JM, Qin X, O'Rourke L, Dimopoulos MA. Daratumumab-based regimens are highly effective and well tolerated in relapsed or refractory multiple myeloma regardless of patient age: subgroup analysis of the phase 3 CASTOR and POLLUX studies. Haematologica. 2020 Jan 31;105(2):468-477. doi: 10.3324/haematol.2019.217448. Print 2020. PMID 31221782
- [Derived] Palumbo A, Chanan-Khan A, Weisel K, Nooka AK, Masszi T, Beksac M, Spicka I, Hungria V, Munder M, Mateos MV, Mark TM, Qi M, Schecter J, Amin H, Qin X, Deraedt W, Ahmadi T, Spencer A, Sonneveld P; CASTOR Investigators. Daratumumab, Bortezomib, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2016 Aug 25;375(8):754-66. doi: 10.1056/NEJMoa1606038. PMID 27557302

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib + Dexamethasone (Vd): Participants received bortezomib 1.3 milligrams per square meter (mg/m^2) subcutaneous (SC) injection on Days 1, 4, 8, and 11 of each 21-day cycle (8 treatment cycles) and dexamethasone 20 milligrams (mg) orally (PO) on Days 1, 2, 4, 5, 8, 9, 11, and 12 of the first 8 bortezomib treatment cycles. Participants who met sponsor confirmed disease progression eligibility criteria received daratumumab monotherapy as a subsequent antimyeloma therapy as follow: daratumumab 16 milligrams per kilogram (mg/kg) intravenous (IV) infusion or daratumumab SC injection (1800 mg fixed dose) weekly for the first 2 cycles, every 2 weeks from Cycle 3 to 6, and then every 4 weeks thereafter.
- Daratumumab + Bortezomib and Dexamethasone (DVd): Participants received daratumumab 16 mg/kg IV infusion weekly or daratumumab SC injection (1800 mg fixed dose) for the first 3 cycles, on Day 1 of Cycles 4-8, and then every 4 weeks thereafter, bortezomib 1.3 mg/m^2 SC injection administration on Days 1, 4, 8, and 11 of each 21-day cycle (8 treatment cycles) and dexamethasone 20 mg orally on Days 1, 2, 4, 5, 8, 9, 11, and 12 of the first 8 bortezomib treatment cycles.
Period: Overall Study
Arm/Group | Bortezomib + Dexamethasone (Vd) | Daratumumab + Bortezomib and Dexamethasone (DVd)
Started | 247 | 251
Daratumumab Monotherapy | 87 | 0
Completed | 0 | 0
Not Completed | 247 | 251
Not completed — Death | 170 | 148
Not completed — Withdrawal by Subject | 19 | 10
Not completed — Lost to Follow-up | 3 | 3
Not completed — Uspecified | 55 | 90

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bortezomib + Dexamethasone (Vd) | Daratumumab + Bortezomib and Dexamethasone (DVd) | Total
Number analyzed (Participants) | 247 | 251 | 498
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (9.81) | 62.8 (9.66) | 63.4 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 114 | 213
  Male | 148 | 137 | 285
Region of Enrollment [Number; unit: participants]
  Australia | 20 | 23 | 43
  Brazil | 9 | 13 | 22
  Czech Republic | 19 | 16 | 35
  Germany | 21 | 21 | 42
  Hungary | 14 | 16 | 30
  Italy | 25 | 24 | 49
  Korea, Republic of | 8 | 10 | 18
  Mexico | 1 | 2 | 3
  Netherlands | 14 | 11 | 25
  Poland | 18 | 16 | 34
  Russian Federation | 13 | 21 | 34
  Spain | 19 | 10 | 29
  Sweden | 9 | 10 | 19
  Turkey | 14 | 14 | 28
  Ukraine | 22 | 28 | 50
  United States | 21 | 16 | 37
Stage of Disease (ISS) [Number; unit: participants] — The International Staging System (ISS) system consists of stage I: beta2-microglobulin less than (<) 3.5 milligrams per liter(mg/L) and albumin greater than or equal to (>=) 3.5 grams (g) per 100 mL; stage II: neither stage I nor stage III and stage III:beta2-microglobulin >= 5.5 mg/L. The higher of staging, the worst of outcome.
  participants
    I | 96 | 98 | 194
    II | 100 | 94 | 194
    III | 51 | 59 | 110
No. of Prior Lines of Therapy [Number; unit: participants]
  1 | 113 | 122 | 235
  2 | 74 | 70 | 144
  3 | 32 | 37 | 69
  >3 | 28 | 22 | 50

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as duration from date of randomization to either progressive disease (PD)/death, whichever occurred first. PD was defined as meeting any one of following criteria: Increase of greater than equal to (>=)25 percent (%) in level of serum M-protein from lowest response value and absolute increase must be >=0.5 gram per deciliter (g/dL); Increase of >=25% in 24-hour urinary light chain excretion (urine M-protein) from lowest response value and absolute increase must be >=200 mg/24hours; Only in participants without measurable serum and urine M-protein levels: increase of >=25% in difference between involved and uninvolved FLC levels from lowest response value and absolute increase must be >10 mg/dL; Definite increase in size of existing bone lesions or soft tissue plasmacytomas; Definite development of new bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder.
Time Frame: From the date of randomization to either progressive disease or death, whichever occurred first (approximately 1 year 4 months)
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bortezomib + Dexamethasone (Vd): Participants received bortezomib 1.3 milligrams per square meter (mg/m^2) subcutaneous (SC) injection on Days 1, 4, 8, and 11 of each 21-day cycle (8 treatment cycles) and dexamethasone 20 milligrams (mg) orally (PO) on Days 1, 2, 4, 5, 8, 9, 11, and 12 of the first 8 bortezomib treatment cycles. Participants who met sponsor-confirmed disease progression eligibility criteria received daratumumab monotherapy as a subsequent antimyeloma therapy as follow: daratumumab 16 milligrams per kilogram (mg/kg) intravenous (IV) infusion or daratumumab SC injection (1800 mg fixed dose) weekly for the first 2 cycles, every 2 weeks from Cycle 3 to 6, and then every 4 weeks thereafter.
Arm/Group | Bortezomib + Dexamethasone (Vd) | Daratumumab + Bortezomib and Dexamethasone (DVd)
Number analyzed (Participants) | 247 | 251
months | 7.16 [6.21 to 7.85] | NA [12.25 to NA] — Median and Upper limit of 95% CI was not estimable due to short follow-up by participants.

2. Secondary Outcome: Time to Disease Progression (TTP)
Description: TTP was defined as time from date of randomization to date of first documented evidence of progressive disease (PD). PD was defined as meeting any one of following criteria: Increase of >=25% in level of serum M-protein from lowest response value and absolute increase must be >=0.5 g/dL; Increase of >=25% in 24-hour urinary light chain excretion (urine M-protein) from lowest response value and absolute increase must be >=200 mg/24hours; Only in participants without measurable serum and urine M-protein levels: increase of >=25% in difference between involved and uninvolved free light chain (FLC) levels from lowest response value and absolute increase must be >10 milligram per deciliter (mg/dL); Definite increase in size of existing bone lesions or soft tissue plasmacytomas; Definite development of new bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to Plasma Cell (PC) proliferative disorder.
Time Frame: From the date of randomization to the date of first documented evidence of progression or death due to PD whichever occurred first (approximately 6 years 9 months)
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib + Dexamethasone (Vd) | Daratumumab + Bortezomib and Dexamethasone (DVd)
Number analyzed (Participants) | 247 | 251
months | 7.29 [6.41 to 8.08] | NA [12.25 to NA] — Median and Upper limit of 95% CI was not estimable due to short follow-up by participants.

3. Secondary Outcome: Percentage of Participants With a Very Good Partial Response (VGPR) or Better
Description: Response rate of VGPR or better was defined as the percentage of participants who achieved VGPR and CR (including sCR) according to the IMWG criteria during or after the study treatment. IMWG criteria for VGPR: Serum and urine M-component detectable by immunofixation but not on electrophoresis, or >=90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours, if the serum and urine M-protein are not measurable, a decrease of >90% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria, in addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas is also required; CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, and <5% PCs in bone marrow; sCR: CR and normal FLC ratio, absence of clonal PCs by immunohistochemistry, immunofluorescence or 2 to 4 color flow cytometry.
Time Frame: Up to disease progression (approximately 6 years 9 months)
Population: The response evaluable analysis set is defined as participants who have a confirmed diagnosis of multiple myeloma and measurable disease at baseline or screening visit, received at least 1 administration of study treatment, and had at least 1 post baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bortezomib + Dexamethasone (Vd) | Daratumumab + Bortezomib and Dexamethasone (DVd)
Number analyzed (Participants) | 234 | 240
percentage of participants | 29.1 [23.3 to 35.3] | 59.2 [52.7 to 65.4]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: The Overall response rate was defined as the percentage of participants who achieved stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) according to the International Myeloma Working Group (IMWG) criteria, during the study or during follow up. IMWG criteria for PR: >=50% reduction of serum M-protein and reduction in 24 hour urinary M-protein by >=90% or to <200 mg/24 hours, if the serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria, in addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: Up to disease progression (approximately 6 years 9 months)
Population: The response-evaluable analysis set is defined as participants who have confirmed diagnosis of multiple myeloma and measurable disease at baseline or screening visit, received at least 1 administration of study treatment and had at least 1 post baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bortezomib + Dexamethasone (Vd) | Daratumumab + Bortezomib and Dexamethasone (DVd)
Number analyzed (Participants) | 234 | 240
percentage of participants | 63.2 [56.7 to 69.4] | 82.9 [77.5 to 87.5]

5. Secondary Outcome: Percentage of Participants With Negative Minimal Residual Disease (MRD)
Description: The Minimal Residual Disease negativity rate was defined as the percentage of participants who had negative MRD assessment at any timepoint after the first dose of study drugs by evaluation of bone marrow aspirates or whole blood. MRD was assessed in participants who achieved complete response or stringent complete response (CR/sCR). IMWG criteria for CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, and <5% PCs in bone marrow; sCR: CR plus normal FLC ratio, absence of clonal PCs by immunohistochemistry, immunofluorescence or 2 to 4 color flow cytometry.
Time Frame: Up to disease progression (approximately 6 years 9 months)
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Bortezomib + Dexamethasone (Vd) | Daratumumab + Bortezomib and Dexamethasone (DVd)
Number analyzed (Participants) | 247 | 251
percentage of participants | 2.8 | 13.5

6. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival was measured from the date of randomization to the date of the participant's death.
Time Frame: Up to 6 years 9 months
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib + Dexamethasone (Vd) | Daratumumab + Bortezomib and Dexamethasone (DVd)
Number analyzed (Participants) | 247 | 251
months | 38.51 [31.18 to 46.23] | 49.58 [42.18 to 62.32]

ADVERSE EVENTS:
Time Frame: Up to 6 years 9 months
Description: Safety population included all randomized participants who had at least 1 administration of any of the study treatment (partial or complete).
Groups:
- Bortezomib + Dexamethasone (Vd): Participants received bortezomib 1.3 milligrams per square meter (mg/m^2) subcutaneous (SC) injection on Days 1, 4, 8, and 11 of each 21-day cycle (8 treatment cycles) and dexamethasone 20 milligrams (mg) orally (PO) on Days 1, 2, 4, 5, 8, 9, 11, and 12 of the first 8 bortezomib treatment cycles.
- Switch From Bortezomib + Dexamethasone (Vd) to Daratumumab Monotherapy: Participants in Vd group, who met sponsor confirmed disease progression eligibility criteria received daratumumab monotherapy as a subsequent antimyeloma therapy as follow: daratumumab 16 milligrams per kilogram (mg/kg) intravenous (IV) infusion or daratumumab SC injection (1800 mg fixed dose) weekly for the first 2 cycles, every 2 weeks from Cycle 3 to 6, and then every 4 weeks thereafter.
Arm/Group | Bortezomib + Dexamethasone (Vd) | Daratumumab + Bortezomib and Dexamethasone (DVd) | Switch From Bortezomib + Dexamethasone (Vd) to Daratumumab Monotherapy
Serious Adverse Events (participants affected / at risk) | 81/237 | 134/243 | 7/87
Other Adverse Events (participants affected / at risk) | 217/237 | 238/243 | 29/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib + Dexamethasone (Vd) (N=237) | Daratumumab + Bortezomib and Dexamethasone (DVd) (N=243) | Switch From Bortezomib + Dexamethasone (Vd) to Daratumumab Monotherapy (N=87)
Anaemia (Blood and lymphatic system disorders) | 1 | 9 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 6 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 2 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 6 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 2 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Age-related macular degeneration (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 3 | 0 | 0
Condition aggravated (General disorders) | 3 | 0 | 0
Fatigue (General disorders) | 0 | 3 | 0
General physical health deterioration (General disorders) | 3 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 4 | 7 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Brain abscess (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 7 | 0
Catheter site infection (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0
Fungal oesophagitis (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 3 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
Haemophilus bacteraemia (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 3 | 0
Influenza (Infections and infestations) | 2 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 2 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Ophthalmic herpes simplex (Infections and infestations) | 1 | 0 | 0
Paraspinal abscess (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 24 | 26 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 2 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1 | 0
Pneumonia serratia (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0
Pulmonary nocardiosis (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 2 | 4 | 0
Septic shock (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 6 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 3 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Electrocardiogram QT interval abnormal (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 3 | 0
Monoparesis (Nervous system disorders) | 1 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 4 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Myeloma cast nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 0 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Gastrointestinal candidiasis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib + Dexamethasone (Vd) (N=237) | Daratumumab + Bortezomib and Dexamethasone (DVd) (N=243) | Switch From Bortezomib + Dexamethasone (Vd) to Daratumumab Monotherapy (N=87)
Anaemia (Blood and lymphatic system disorders) | 75 | 68 | 1
Leukopenia (Blood and lymphatic system disorders) | 12 | 23 | 0
Lymphopenia (Blood and lymphatic system disorders) | 9 | 33 | 0
Neutropenia (Blood and lymphatic system disorders) | 23 | 47 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 105 | 145 | 0
Abdominal pain (Gastrointestinal disorders) | 10 | 14 | 0
Abdominal pain upper (Gastrointestinal disorders) | 7 | 19 | 0
Constipation (Gastrointestinal disorders) | 37 | 56 | 0
Diarrhoea (Gastrointestinal disorders) | 53 | 88 | 0
Dyspepsia (Gastrointestinal disorders) | 13 | 9 | 0
Nausea (Gastrointestinal disorders) | 27 | 37 | 2
Vomiting (Gastrointestinal disorders) | 9 | 30 | 0
Asthenia (General disorders) | 36 | 27 | 0
Fatigue (General disorders) | 58 | 57 | 0
Oedema (General disorders) | 9 | 13 | 0
Oedema peripheral (General disorders) | 20 | 48 | 0
Pyrexia (General disorders) | 26 | 42 | 1
Bronchitis (Infections and infestations) | 14 | 35 | 1
Conjunctivitis (Infections and infestations) | 8 | 26 | 0
Herpes zoster (Infections and infestations) | 5 | 17 | 0
Influenza (Infections and infestations) | 6 | 17 | 0
Nasopharyngitis (Infections and infestations) | 9 | 33 | 0
Pneumonia (Infections and infestations) | 9 | 22 | 2
Upper respiratory tract infection (Infections and infestations) | 41 | 88 | 1
Urinary tract infection (Infections and infestations) | 5 | 21 | 0
Alanine aminotransferase increased (Investigations) | 10 | 20 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 15 | 0
Weight decreased (Investigations) | 3 | 19 | 0
Decreased appetite (Metabolism and nutrition disorders) | 12 | 28 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 17 | 22 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 11 | 17 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 26 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 17 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 48 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 52 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 13 | 21 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 25 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 25 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 15 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 33 | 0
Dizziness (Nervous system disorders) | 25 | 31 | 0
Headache (Nervous system disorders) | 14 | 29 | 0
Neuralgia (Nervous system disorders) | 26 | 34 | 0
Paraesthesia (Nervous system disorders) | 14 | 13 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 90 | 122 | 0
Insomnia (Psychiatric disorders) | 36 | 44 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 23 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 71 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 47 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 12 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 14 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 13 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 13 | 3
Rash (Skin and subcutaneous tissue disorders) | 7 | 16 | 0
Hypertension (Vascular disorders) | 8 | 30 | 2
Hypotension (Vascular disorders) | 10 | 13 | 2
Chills (General disorders) | 3 | 12 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.